CLINICAL TRIAL: NCT02748330
Title: A Randomized, Open-label, Active-controlled, Parallel-group Study to Investigate the Platelet Inhibition of Ticagrelor Versus Clopidogrel in Patients With Stable Coronary Artery Disease and Type 2 Diabetes Mellitus After Recent Elective Percutaneous Coronary Intervention
Brief Title: Platelet Inhibition of Ticagrelor Versus Clopidogrel in Type 2 Diabetic Patients After Elective Percutaneous Coronary Intervention
Acronym: PLATIDE-PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-873; ESR-14-10403 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Oral ticagrelor 90 mg tablet, twice daily for 15±2 days. Oral aspirin 100 mg tablet, once daily for 15±2 days
  Interventions: Drug: Ticagrelor; Drug: Aspirin
- Clopidogrel (Active Comparator): Oral clopidogrel 75 mg tablet, once daily for 15±2 days. Oral aspirin 100 mg tablet, once daily for 15±2 days
  Interventions: Drug: Clopidogrel; Drug: Aspirin

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Clopidogrel — Clopidogrel
  Other Names: Plavix
  Arms: Clopidogrel
Drug: Aspirin — Acetylsalicylic acid

SUMMARY:
This will be a single-center, randomized, open-label, active-controlled, parallel-group study to investigate the platelet inhibition of Ticagrelor versus Clopidogrel with acetylsalicylic acid (ASA) as background therapy in approximate 40 patients with stable coronary artery disease (SCAD) and type 2 diabetes mellitus (DM) after recent successful elective percutaneous coronary intervention (PCI) by evaluation of the P2Y12 reaction unit (PRU) by VerifyNow P2Y12 assay at 2-4 hours after the first study drug dose on treatment day 15±2.

DETAILED DESCRIPTION:
The study will consist of a screening period, a 15±2 day treatment period, and a 7 day follow-up period. The screening period will be up to 7 days. Once each patient has signed the informed consent, the eligibility of the patient will be determined at screening, and laboratory assessments will be taken (Visit 1). During the treatment period, patients participating in the study will be randomized to receive either Ticagrelor with ASA, or Clopidogrel with ASA for 15±2 days. The final dose of study medication will be administered at the study site in the morning of day 15±2. Study visits at the beginning (Visit 2) and the end of the treatment period (Visit 4) will allow assessment of platelet function. At 7±1 days after Visit 2, a telephone visit (Visit 3) will be carried out for collection of information on concomitant medication, adverse events (including vascular events), and safety end point events. After the platelet function tests at Visit 4 are finished, patients in both groups will discontinue their study medication (end of treatment, EOT). A follow-up period will begin at 1 day after Visit 4 and continue for 7 days. During the follow-up period, patients in Ticagrelor group will take Clopidogrel 600 mg loading dose on the first day, followed by Clopidogrel 75 mg maintenance dose from the second day for 6 days; patients in Clopidogrel group will continue taking Clopidogrel 75 mg maintenance dose for 7 days. Both adverse events (including vascular events) and safety end point events will be collected at the safety visit (Visit 5), which will occur 7 days after Visit 4. The study will last approximately 4 weeks per patient. After the informed consents are signed by the patients, all adverse events (including vascular events), safety end point events and concomitant medications will be recorded at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent (by patient or appropriate designee according to local regulations) prior to any study specific procedures.
2. Aged 18 years or older, male or female.
3. Documented stable coronary artery disease (CAD) fulfilling any of the following:

   * History of stable angina pectoris with angiographic evidence of CAD (diameter stenosis ≥ 50%) in major, i.e., left main, left anterior descending, left circumflex, and right coronary arteries.
   * History of previous myocardial infarction (MI)
   * History of coronary revascularization, i.e., percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG), not including the elective PCI during the index hospitalization
4. Documented history of type 2 diabetes mellitus.
5. At least 24 hours after but within 14 days of angiographically successful elective PCI without complications.

   * Post-procedural residual diameter stenosis of the treated lesions < 20% in patients with stent implantation or < 50% in those with balloon angioplasty
   * Post-procedural thrombolysis in myocardial infarction (TIMI) grade 3 flow in treated vessels
6. Negative cardiac troponin test before the index elective PCI.
7. Taking Clopidogrel 75 mg daily dose for at least 7 days or taking Clopidogrel 75 mg daily dose for less than 7 days but with 300 to 600 mg Clopidogrel loading dose before PCI.
8. Taking acetylsalicylic acid (ASA) 100 mg daily treatment for at least 7 days or taking ASA 100 mg daily dose for less than 7 days but with 300 mg ASA loading dose before PCI.
9. Females with childbearing potential (i.e., females who are not post-menopausal or surgically sterile) must:

   * have a negative urine or blood pregnancy test at enrolment and prior to randomization;
   * currently be using a hormonal contraceptive and agree to continue its use in addition to using double-barrier local contraception (i.e., intra-uterine device plus spermicidal and condom for male partner) from screening through study completion.

Exclusion Criteria:

1. Patients who had acute coronary syndrome (ACS) within 12 months of screening.
2. Occurrence of myocardial infarction (MI) related to index elective PCI (type 4a MI) or myocardial infarction related to stent thrombosis (type 4b MI) according to the Third Universal Definition of Myocardial Infarction.
3. Use of parenteral antithrombotic agents, e.g., glycoprotein IIb/IIIa inhibitors (GPIs), bivalirudin, unfractionated heparin, enoxaparin or fondaparinux within 24 hours of screening.
4. Use of any oral antithrombotic agents, with the exception of Clopidogrel and ASA, within 30 days of screening.
5. Any other indications (e.g., atrial fibrillation, prosthetic heart valve, venous thromboembolism, ventricular thrombosis, et al) for antithrombotic treatment other than ASA 100 mg daily, Clopidogrel and Ticagrelor during study period.
6. Concomitant therapy with moderate or strong cytochrome P-450 (CYP) 3A inhibitors, CYP 3A substrates with narrow therapeutic index, or strong CYP 3A inducers during study period.
7. Concomitant therapy with moderate or strong CYP 2C19 inhibitors, CYP 2C19 substrates with narrow therapeutic index, or strong CYP 2C19 inducers during study period.
8. Increased bleeding risk including:

   * recent (within 30 days of screening) gastrointestinal (GI) bleeding;
   * any history of intracranial, intraocular, retroperitoneal, or spinal bleeding;
   * recent (within 30 days of screening) major trauma or major surgery;
   * sustained uncontrolled hypertension (systolic blood pressure [SBP] > 180 mmHg or diastolic blood pressure [DBP] > 100 mmHg);
   * history of hemorrhagic disorders that can increase the risk of bleeding, e.g., haemophilia, von Willebrand's disease;
   * inability to discontinue required concomitant therapy with non-selective non-steroidal anti-inflammatory drugs (NSAIDs) at screening;
   * platelet count less than 100,000/mm3 or hemoglobin < 10 g/dL.
9. Contraindication or other reason that ASA, Clopidogrel, or Ticagrelor should not be administered (e.g., hypersensitivity, active bleeding [including active pathological bleeding], any bleeding tendency [coagulation defects], moderate and severe hepatic impairment, risk of bradycardia, chronic obstructive pulmonary disease, chronic or active asthma, hyperuricemia, gout, etc.).
10. History of intolerance to ASA, Clopidogrel or Ticagrelor.
11. Patients that are scheduled for CABG during the study period.
12. Patient requires dialysis or has a creatinine clearance (Clcr) < 30 mL/min as calculated by the Cockcroft-Gault equation: Clcr = (140 - Age) × WT / (72 × Scr) (× 0.85 for females), where WT is weight in kg, Scr is serum creatinine in mg/dL.
13. Any acute or chronic unstable conditions in the past 30 days or other conditions which, in the opinion of the investigator, may either put the patient at risk or influence the result of the study (e.g., active cancer, risk for non-compliance, risk for being lost to follow-up).
14. Participation in another investigational drug or device study within 30 days of screening.
15. Involvement in the planning and conduct of the study (applies to investigators, contract research organization staff, and study site staff).
16. History of drug addiction or alcohol abuse in the previous 2 years.
17. Recent (within 30 days of screening) blood donation.
18. Known pregnancy, breast-feeding, or intend to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
P2Y12 reaction unit (PRU) | 15±2 days
  The PRU by VerifyNow P2Y12 assay at 2-4 hours after the first study drug dose on day 15±2

SECONDARY OUTCOMES:
P2Y12 reaction unit (PRU) (before) | 15±2 days
  The PRU by VerifyNow P2Y12 assay before the first study drug dose on day 15±2
Percent inhibition (% Inhibition) | 15±2 days
  The % Inhibition by VerifyNow P2Y12 assay at 2-4 hours after the first study drug dose on day 15±2
Percent inhibition (% Inhibition) (before) | 15±2 days
  The % Inhibition by VerifyNow P2Y12 assay before the first study drug dose on day 15±2
High on-treatment platelet reactivity (HOPR) | 15±2 days
  The rate of HOPR by VerifyNow P2Y12 assay at 2-4 hours after the first study drug dose on day 15±2
High on-treatment platelet reactivity (HOPR) (before) | 15±2 days
  The rate of HOPR by VerifyNow P2Y12 assay before the first study drug dose on day 15±2
Non-coronary artery bypass graft (CABG) related major bleeding | 15±2 days
  The rate of non-CABG related major bleeding according to Platelet Inhibition and Patient Outcome (PLATO) study definition up to day 15±2.
Non-coronary artery bypass graft (CABG) related major or minor bleeding | 15±2 days
  The rate of non-CABG related major or minor bleeding according to PLATO definition up to day 15±2.
Non-coronary artery bypass graft (CABG) related major or minor or minimal bleeding | 15±2 days
  The rate of non-CABG related major or minor or minimal bleeding according to PLATO definition up to day 15±2.

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Angiolillo DJ, Fernandez-Ortiz A, Bernardo E, Ramirez C, Sabate M, Jimenez-Quevedo P, Hernandez R, Moreno R, Escaned J, Alfonso F, Banuelos C, Costa MA, Bass TA, Macaya C. Platelet function profiles in patients with type 2 diabetes and coronary artery disease on combined aspirin and clopidogrel treatment. Diabetes. 2005 Aug;54(8):2430-5. doi: 10.2337/diabetes.54.8.2430. PMID 16046311
- [Result] Angiolillo DJ, Bernardo E, Sabate M, Jimenez-Quevedo P, Costa MA, Palazuelos J, Hernandez-Antolin R, Moreno R, Escaned J, Alfonso F, Banuelos C, Guzman LA, Bass TA, Macaya C, Fernandez-Ortiz A. Impact of platelet reactivity on cardiovascular outcomes in patients with type 2 diabetes mellitus and coronary artery disease. J Am Coll Cardiol. 2007 Oct 16;50(16):1541-7. doi: 10.1016/j.jacc.2007.05.049. Epub 2007 Oct 1. PMID 17936152
- [Result] Angiolillo DJ, Fernandez-Ortiz A, Bernardo E, Alfonso F, Macaya C, Bass TA, Costa MA. Variability in individual responsiveness to clopidogrel: clinical implications, management, and future perspectives. J Am Coll Cardiol. 2007 Apr 10;49(14):1505-16. doi: 10.1016/j.jacc.2006.11.044. Epub 2007 Mar 26. PMID 17418288
- [Result] Angiolillo DJ, Shoemaker SB, Desai B, Yuan H, Charlton RK, Bernardo E, Zenni MM, Guzman LA, Bass TA, Costa MA. Randomized comparison of a high clopidogrel maintenance dose in patients with diabetes mellitus and coronary artery disease: results of the Optimizing Antiplatelet Therapy in Diabetes Mellitus (OPTIMUS) study. Circulation. 2007 Feb 13;115(6):708-16. doi: 10.1161/CIRCULATIONAHA.106.667741. Epub 2007 Jan 29. PMID 17261652
- [Result] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Result] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214
- [Result] Arnold SV, Morrow DA, Lei Y, Cohen DJ, Mahoney EM, Braunwald E, Chan PS. Economic impact of angina after an acute coronary syndrome: insights from the MERLIN-TIMI 36 trial. Circ Cardiovasc Qual Outcomes. 2009 Jul;2(4):344-53. doi: 10.1161/CIRCOUTCOMES.108.829523. Epub 2009 Jun 2. PMID 20031860
- [Result] Beckman JA, Creager MA, Libby P. Diabetes and atherosclerosis: epidemiology, pathophysiology, and management. JAMA. 2002 May 15;287(19):2570-81. doi: 10.1001/jama.287.19.2570. PMID 12020339
- [Result] Caiazzo G, De Rosa S, Torella D, Spaccarotella C, Mongiardo A, Giampa S, Micieli M, Palella E, Gulletta E, Indolfi C. Administration of a loading dose has no additive effect on platelet aggregation during the switch from ongoing clopidogrel treatment to ticagrelor in patients with acute coronary syndrome. Circ Cardiovasc Interv. 2014 Feb;7(1):104-12. doi: 10.1161/CIRCINTERVENTIONS.113.000512. Epub 2014 Jan 21. PMID 24449597
- [Result] Cannon CP, Harrington RA, James S, Ardissino D, Becker RC, Emanuelsson H, Husted S, Katus H, Keltai M, Khurmi NS, Kontny F, Lewis BS, Steg PG, Storey RF, Wojdyla D, Wallentin L; PLATelet inhibition and patient Outcomes Investigators. Comparison of ticagrelor with clopidogrel in patients with a planned invasive strategy for acute coronary syndromes (PLATO): a randomised double-blind study. Lancet. 2010 Jan 23;375(9711):283-93. doi: 10.1016/S0140-6736(09)62191-7. Epub 2010 Jan 13. PMID 20079528
- [Result] Colwell JA, Nesto RW. The platelet in diabetes: focus on prevention of ischemic events. Diabetes Care. 2003 Jul;26(7):2181-8. doi: 10.2337/diacare.26.7.2181. PMID 12832332
- [Result] Creager MA, Luscher TF, Cosentino F, Beckman JA. Diabetes and vascular disease: pathophysiology, clinical consequences, and medical therapy: Part I. Circulation. 2003 Sep 23;108(12):1527-32. doi: 10.1161/01.CIR.0000091257.27563.32. No abstract available. PMID 14504252
- [Result] Davies SL. Ticagrelor. Drugs Today (Barc). 2010 Apr;46(4):243-50. doi: 10.1358/dot.2010.46.4.1467168. PMID 20502721
- [Result] Diodati JG, Saucedo JF, French JK, Fung AY, Cardillo TE, Henneges C, Effron MB, Fisher HN, Angiolillo DJ. Effect on platelet reactivity from a prasugrel loading dose after a clopidogrel loading dose compared with a prasugrel loading dose alone: Transferring From Clopidogrel Loading Dose to Prasugrel Loading Dose in Acute Coronary Syndrome Patients (TRIPLET): a randomized controlled trial. Circ Cardiovasc Interv. 2013 Oct 1;6(5):567-74. doi: 10.1161/CIRCINTERVENTIONS.112.000063. Epub 2013 Sep 24. PMID 24065443
- [Result] Ferreira IA, Eybrechts KL, Mocking AI, Kroner C, Akkerman JW. IRS-1 mediates inhibition of Ca2+ mobilization by insulin via the inhibitory G-protein Gi. J Biol Chem. 2004 Jan 30;279(5):3254-64. doi: 10.1074/jbc.M305474200. Epub 2003 Nov 5. PMID 14602724
- [Result] Ferreira IA, Mocking AI, Feijge MA, Gorter G, van Haeften TW, Heemskerk JW, Akkerman JW. Platelet inhibition by insulin is absent in type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2006 Feb;26(2):417-22. doi: 10.1161/01.ATV.0000199519.37089.a0. Epub 2005 Dec 8. PMID 16339499
- [Result] Fuster V, Stein B, Ambrose JA, Badimon L, Badimon JJ, Chesebro JH. Atherosclerotic plaque rupture and thrombosis. Evolving concepts. Circulation. 1990 Sep;82(3 Suppl):II47-59. PMID 2203564
- [Result] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Result] Gurbel PA, Bliden KP, Samara W, Yoho JA, Hayes K, Fissha MZ, Tantry US. Clopidogrel effect on platelet reactivity in patients with stent thrombosis: results of the CREST Study. J Am Coll Cardiol. 2005 Nov 15;46(10):1827-32. doi: 10.1016/j.jacc.2005.07.056. Epub 2005 Oct 19. PMID 16286166
- [Result] Gurbel PA, Tantry US. Clopidogrel resistance? Thromb Res. 2007;120(3):311-21. doi: 10.1016/j.thromres.2006.08.012. Epub 2006 Nov 14. PMID 17109936
- [Result] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Result] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878
- [Result] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301
- [Result] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Result] Hemingway H, McCallum A, Shipley M, Manderbacka K, Martikainen P, Keskimaki I. Incidence and prognostic implications of stable angina pectoris among women and men. JAMA. 2006 Mar 22;295(12):1404-11. doi: 10.1001/jama.295.12.1404. PMID 16551712
- [Result] Husted S, Emanuelsson H, Heptinstall S, Sandset PM, Wickens M, Peters G. Pharmacodynamics, pharmacokinetics, and safety of the oral reversible P2Y12 antagonist AZD6140 with aspirin in patients with atherosclerosis: a double-blind comparison to clopidogrel with aspirin. Eur Heart J. 2006 May;27(9):1038-47. doi: 10.1093/eurheartj/ehi754. Epub 2006 Feb 13. PMID 16476694
- [Result] Husted S. Unmet needs in oral antiplatelet therapy with ADP receptor blocking agents. Fundam Clin Pharmacol. 2009 Feb;23(1):1-9. doi: 10.1111/j.1472-8206.2008.00660.x. PMID 19267766
- [Result] James S, Angiolillo DJ, Cornel JH, Erlinge D, Husted S, Kontny F, Maya J, Nicolau JC, Spinar J, Storey RF, Stevens SR, Wallentin L; PLATO Study Group. Ticagrelor vs. clopidogrel in patients with acute coronary syndromes and diabetes: a substudy from the PLATelet inhibition and patient Outcomes (PLATO) trial. Eur Heart J. 2010 Dec;31(24):3006-16. doi: 10.1093/eurheartj/ehq325. Epub 2010 Aug 29. PMID 20802246
- [Result] Javitz HS, Ward MM, Watson JB, Jaana M. Cost of illness of chronic angina. Am J Manag Care. 2004 Oct;10(11 Suppl):S358-69. PMID 15603245
- [Result] Jneid H, Anderson JL, Wright RS, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP. 2012 ACCF/AHA focused update of the guideline for the management of patients with unstable angina/non-ST-elevation myocardial infarction (updating the 2007 guideline and replacing the 2011 focused update): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2012 Aug 14;60(7):645-81. doi: 10.1016/j.jacc.2012.06.004. Epub 2012 Jul 16. No abstract available. PMID 22809746
- [Result] Judge HM, Buckland RJ, Sugidachi A, Jakubowski JA, Storey RF. The active metabolite of prasugrel effectively blocks the platelet P2Y12 receptor and inhibits procoagulant and pro-inflammatory platelet responses. Platelets. 2008 Mar;19(2):125-33. doi: 10.1080/09537100701694144. PMID 18297550
- [Result] Kowalczyk M, Banach M, Mikhailidis DP, Hannam S, Rysz J. Ticagrelor--a new platelet aggregation inhibitor in patients with acute coronary syndromes. An improvement of other inhibitors? Med Sci Monit. 2009 Dec;15(12):MS24-30. PMID 19946242
- [Result] Leal J, Luengo-Fernandez R, Gray A, Petersen S, Rayner M. Economic burden of cardiovascular diseases in the enlarged European Union. Eur Heart J. 2006 Jul;27(13):1610-9. doi: 10.1093/eurheartj/ehi733. Epub 2006 Feb 22. PMID 16495286
- [Result] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Result] Luscher TF, Creager MA, Beckman JA, Cosentino F. Diabetes and vascular disease: pathophysiology, clinical consequences, and medical therapy: Part II. Circulation. 2003 Sep 30;108(13):1655-61. doi: 10.1161/01.CIR.0000089189.70578.E2. No abstract available. PMID 14517152
- [Result] Maddox TM, Reid KJ, Spertus JA, Mittleman M, Krumholz HM, Parashar S, Ho PM, Rumsfeld JS. Angina at 1 year after myocardial infarction: prevalence and associated findings. Arch Intern Med. 2008 Jun 23;168(12):1310-6. doi: 10.1001/archinte.168.12.1310. PMID 18574088
- [Result] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Result] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Result] Murray CJ, Lopez AD. Alternative projections of mortality and disability by cause 1990-2020: Global Burden of Disease Study. Lancet. 1997 May 24;349(9064):1498-504. doi: 10.1016/S0140-6736(96)07492-2. PMID 9167458
- [Result] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Result] Schneider DJ. Factors contributing to increased platelet reactivity in people with diabetes. Diabetes Care. 2009 Apr;32(4):525-7. doi: 10.2337/dc08-1865. No abstract available. PMID 19336636
- [Result] Scirica BM, Cannon CP, Emanuelsson H, Michelson EL, Harrington RA, Husted S, James S, Katus H, Pais P, Raev D, Spinar J, Steg PG, Storey RF, Wallentin L; PLATO Investigators. The incidence of bradyarrhythmias and clinical bradyarrhythmic events in patients with acute coronary syndromes treated with ticagrelor or clopidogrel in the PLATO (Platelet Inhibition and Patient Outcomes) trial: results of the continuous electrocardiographic assessment substudy. J Am Coll Cardiol. 2011 May 10;57(19):1908-16. doi: 10.1016/j.jacc.2010.11.056. PMID 21545948
- [Result] Simpson SH, Abdelmoneim AS, Omran D, Featherstone TR. Prevalence of high on-treatment platelet reactivity in diabetic patients treated with aspirin. Am J Med. 2014 Jan;127(1):95.e1-9. doi: 10.1016/j.amjmed.2013.09.019. Epub 2013 Oct 8. PMID 24384107
- [Result] Spertus JA, Salisbury AC, Jones PG, Conaway DG, Thompson RC. Predictors of quality-of-life benefit after percutaneous coronary intervention. Circulation. 2004 Dec 21;110(25):3789-94. doi: 10.1161/01.CIR.0000150392.70749.C7. Epub 2004 Dec 13. PMID 15596563
- [Result] Stefanini GG, Holmes DR Jr. Drug-eluting coronary-artery stents. N Engl J Med. 2013 Jan 17;368(3):254-65. doi: 10.1056/NEJMra1210816. No abstract available. PMID 23323902
- [Result] Steg PG, Bhatt DL, Wilson PW, D'Agostino R Sr, Ohman EM, Rother J, Liau CS, Hirsch AT, Mas JL, Ikeda Y, Pencina MJ, Goto S; REACH Registry Investigators. One-year cardiovascular event rates in outpatients with atherothrombosis. JAMA. 2007 Mar 21;297(11):1197-206. doi: 10.1001/jama.297.11.1197. PMID 17374814
- [Result] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Result] Steinhubl SR, Berger PB, Mann JT 3rd, Fry ET, DeLago A, Wilmer C, Topol EJ; CREDO Investigators. Clopidogrel for the Reduction of Events During Observation. Early and sustained dual oral antiplatelet therapy following percutaneous coronary intervention: a randomized controlled trial. JAMA. 2002 Nov 20;288(19):2411-20. doi: 10.1001/jama.288.19.2411. PMID 12435254
- [Result] Stone GW, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Gurbel PA, Xu K, Parise H, Kirtane AJ, Brodie BR, Mehran R, Stuckey TD; ADAPT-DES Investigators. Platelet reactivity and clinical outcomes after coronary artery implantation of drug-eluting stents (ADAPT-DES): a prospective multicentre registry study. Lancet. 2013 Aug 17;382(9892):614-23. doi: 10.1016/S0140-6736(13)61170-8. Epub 2013 Jul 26. PMID 23890998
- [Result] Storey RF, Husted S, Harrington RA, Heptinstall S, Wilcox RG, Peters G, Wickens M, Emanuelsson H, Gurbel P, Grande P, Cannon CP. Inhibition of platelet aggregation by AZD6140, a reversible oral P2Y12 receptor antagonist, compared with clopidogrel in patients with acute coronary syndromes. J Am Coll Cardiol. 2007 Nov 6;50(19):1852-6. doi: 10.1016/j.jacc.2007.07.058. Epub 2007 Oct 23. PMID 17980251
- [Result] Storey RF, Angiolillo DJ, Patil SB, Desai B, Ecob R, Husted S, Emanuelsson H, Cannon CP, Becker RC, Wallentin L. Inhibitory effects of ticagrelor compared with clopidogrel on platelet function in patients with acute coronary syndromes: the PLATO (PLATelet inhibition and patient Outcomes) PLATELET substudy. J Am Coll Cardiol. 2010 Oct 26;56(18):1456-62. doi: 10.1016/j.jacc.2010.03.100. PMID 20832963
- [Result] Storey RF, Becker RC, Harrington RA, Husted S, James SK, Cools F, Steg PG, Khurmi NS, Emanuelsson H, Lim ST, Cannon CP, Katus HA, Wallentin L. Pulmonary function in patients with acute coronary syndrome treated with ticagrelor or clopidogrel (from the Platelet Inhibition and Patient Outcomes [PLATO] pulmonary function substudy). Am J Cardiol. 2011 Dec 1;108(11):1542-6. doi: 10.1016/j.amjcard.2011.07.015. Epub 2011 Sep 3. PMID 21890085
- [Result] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Result] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Result] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503